CLINICAL TRIAL: NCT06779643
Title: Efficacy and Safety of Liposomal Bupivacaine and Ropivacaine in Upper Limb Surgery: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Liposomal Bupivacaine and Ropivacaine in Upper Limb Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaguang Duan (Other)
Responsible Party: Sponsor-Investigator, Xiaguang Duan, Deputy Chief of Anesthesiology, Inner Mongolia Baogang Hospital
Organization: Inner Mongolia Baogang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-MER-319
Record Dates: First submitted 2025-01-13; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Upper Limb Injury
MeSH Terms: conditions — Arm Injuries | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- GA group (Experimental): General anesthesia group. Anesthesia induction will be achieved using propofol (1.5-2 mg/kg i.v.), rocuronium (1-2 mg/kg i.v.), and fentanyl (1-2 μg/kg i.v.). Anesthesia will be maintained using sevoflurane or desflurane, with inhaled concentration adjusted based on Bispectral Index (BIS) monitoring. A continuous infusion of remifentanil (0.05-0.2 μg/kg/min) will be administered, with adjustments to maintain blood pressure and heart rate within ±20% of baseline values. Following induction, patients will be mechanically ventilated in pressure-regulated volume control (PRVC) mode. The ventilator (Aestiva; GE Healthcare, Waukesha, Wisconsin, USA) settings will be: tidal volume 6-8 mL/kg, positive end-expiratory pressure 0 cm H2O, inspiratory to expiratory ratio 1:2, respiratory rate 16 breaths per minute (BPM), and fraction of inspired oxygen 41%.
  Interventions: Device: General Anesthesia (GA)
- CBPB group (Experimental): Patients were positioned supine with the head slightly turned to the contralateral side to expose the supraclavicular fossa. The injection site was prepared using standard aseptic techniques. Under ultrasound guidance, a needle was advanced to the vicinity of the brachial plexus. Aspiration was performed to confirm the absence of blood return before the slow, incremental injection of either liposomal bupivacaine [adult dose: 133 mg (10 mL) to 266 mg (20 mL)] or ropivacaine [adult dose: 20 mL of 0.5% ropivacaine, administered via continuous infusion at a rate of 5-10 mL/h; pediatric dose: 0.1% ropivacaine at 0.1-0.2 mL/kg, administered via continuous infusion at 0.05-0.15 mL/kg/h]. Patient responses were closely monitored throughout the procedure.
  Interventions: Device: General Anesthesia (GA); Device: Continuous Brachial Plexus Block

INTERVENTIONS:
Device: General Anesthesia (GA) — Anesthesia induction will be achieved using propofol (1.5-2 mg/kg i.v.), rocuronium (1-2 mg/kg i.v.), and fentanyl (1-2 μg/kg i.v.). Anesthesia will be maintained using sevoflurane or desflurane, with inhaled concentration adjusted based on Bispectral Index (BIS) monitoring. A continuous infusion of remifentanil (0.05-0.2 μg/kg/min) will be administered, with adjustments to maintain blood pressure and heart rate within ±20% of baseline values. Following induction, patients will be mechanically ventilated in pressure-regulated volume control (PRVC) mode. The ventilator (Aestiva; GE Healthcare, Waukesha, Wisconsin, USA) settings will be: tidal volume 6-8 mL/kg, positive end-expiratory pressure 0 cm H2O, inspiratory to expiratory ratio 1:2, respiratory rate 16 breaths per minute (BPM), and fraction of inspired oxygen 41%.
Device: Continuous Brachial Plexus Block — Patients were positioned supine with the head slightly turned to the contralateral side to expose the supraclavicular fossa. The injection site was prepared using standard aseptic techniques. Under ultrasound guidance, a needle was advanced to the vicinity of the brachial plexus. Aspiration was performed to confirm the absence of blood return before the slow, incremental injection of either liposomal bupivacaine [adult dose: 133 mg (10 mL) to 266 mg (20 mL)] or ropivacaine [adult dose: 20 mL of 0.5% ropivacaine, administered via continuous infusion at a rate of 5-10 mL/h; pediatric dose: 0.1% ropivacaine at 0.1-0.2 mL/kg, administered via continuous infusion at 0.05-0.15 mL/kg/h]. Patient responses were closely monitored throughout the procedure.
  Arms: CBPB group

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of liposomal bupivacaine and ropivacaine when used in different brachial plexus blocks and epidural anesthesia for the management of pain associated with burn injuries, digital replantation, and upper limb fractures (including radial, ulnar, humeral, and carpal fractures), as well as hand fractures (including phalangeal and metacarpal fractures). The primary objective is to determine whether liposomal bupivacaine or ropivacaine reduces the required postoperative analgesic dosage in these patient populations.

Specifically, this study will compare brachial plexus blockade with either liposomal bupivacaine or ropivacaine, combined with general anesthesia, against general anesthesia alone to assess the effectiveness of these two local anesthetics in achieving postoperative analgesia.

Enrolled participants will be randomized to one of two treatment arms: either brachial plexus block followed by endotracheal intubation and general anesthesia or general anesthesia alone. Postoperative vital signs, analgesic requirements, and recovery parameters will be continuously monitored and recorded.

DETAILED DESCRIPTION:
Study Design: This study employed a prospective, randomized, comparative, and double-blinded design to assess the superiority and non-inferiority of brachial plexus blockade combined with general anesthesia versus general anesthesia alone for postoperative analgesia in patients with upper limb injuries. Patient recruitment was conducted at Baogang Hospital, Inner Mongolia. This study was approved by the Medical Ethics Committee of Baogang Hospital, Inner Mongolia, and adhered to the principles of the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) guidelines. All participants provided informed consent prior to enrollment.

Patients: Sixty patients aged two years or older with American Society of Anesthesiologists (ASA) physical status classifications I to III, scheduled for surgery due to upper limb injuries between February 2025 and May 2025, were enrolled in this study. Participants were randomly assigned to one of two groups, each containing 30 patients, receiving either brachial plexus blockade combined with general anesthesia or general anesthesia alone.

Randomization and Blinding：This study employed block randomization to generate the random allocation sequence. A block size of 6 was set, and the random sequence was generated using dedicated software (the blockrand package in R version 4.3.2). The allocation of the random sequence was performed by an independent third party, and allocation concealment was implemented using sequentially numbered, sealed, opaque envelopes. The research team remained blinded throughout the randomization process and was not involved in the generation or allocation of the random sequence.

Intervention：Upon arrival to the operating room, patients will be monitored with electrocardiography, blood pressure, and pulse oximetry. Patients will be placed in the prone position with their arms abducted and internally rotated. Ultrasound guidance will be used for all regional anesthesia procedures (SonoSite Edge II; Fujifilm SonoSite, Bothell, WA, USA) with a linear 13-6 MHz ultrasound probe (HFL50x; Fujifilm SonoSite, Bothell, WA, USA). For each block, a 5 mL test dose will be injected initially, followed by observation for clinical signs of a successful block. After confirming correct placement, the remaining dose of the anesthetic agent will be injected. Following administration of the regional anesthesia, general anesthesia with endotracheal intubation will be performed. Anesthesia induction will be achieved using propofol (1.5-2 mg/kg i.v.), rocuronium (1-2 mg/kg i.v.), and fentanyl (1-2 μg/kg i.v.). Anesthesia will be maintained using sevoflurane or desflurane, with inhaled concentration adjusted based on Bispectral Index (BIS) monitoring. A continuous infusion of remifentanil (0.05-0.2 μg/kg/min) will be administered, with adjustments to maintain blood pressure and heart rate within ±20% of baseline values. Following induction, patients will be mechanically ventilated in pressure-regulated volume control (PRVC) mode. The ventilator (Aestiva; GE Healthcare, Waukesha, Wisconsin, USA) settings will be: tidal volume 6-8 mL/kg, positive end-expiratory pressure 0 cm H2O, inspiratory to expiratory ratio 1:2, respiratory rate 16 breaths per minute (BPM), and fraction of inspired oxygen 41%.

Continuous Brachial Plexus Block Procedure: Patients were positioned supine with the head slightly turned to the contralateral side to expose the supraclavicular fossa. The injection site was prepared using standard aseptic techniques. Under ultrasound guidance, a needle was advanced to the vicinity of the brachial plexus. Aspiration was performed to confirm the absence of blood return before the slow, incremental injection of either liposomal bupivacaine [adult dose: 133 mg (10 mL) to 266 mg (20 mL)] or ropivacaine [adult dose: 20 mL of 0.5% ropivacaine, administered via continuous infusion at a rate of 5-10 mL/h; pediatric dose: 0.1% ropivacaine at 0.1-0.2 mL/kg, administered via continuous infusion at 0.05-0.15 mL/kg/h]. Patient responses were closely monitored throughout the procedure.

Outcomes and Measures: Postoperative assessments were conducted in the ward by two nurses blinded to group assignment and specifically trained in the study protocols. These nurses performed in-person evaluations at the following time points: pre-treatment (baseline), and then postoperatively at 2 hours, 6 hours, 12 hours, and 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age: Two years or older.
* ASA Physical Status: American Society of Anesthesiologists (ASA) physical status classification of I, II, or III.
* Surgical Indication: Patients requiring surgical treatment for any of the following upper limb injuries: Burn injuries. Digital replantation. Upper limb fractures, including fractures of the radius, ulna, humerus, and carpal bones. Hand fractures, including fractures of the phalanges and metacarpals.
* Patients scheduled to undergo either a continuous brachial plexus block combined with general anesthesia or general anesthesia alone.
* Patients (or their legal guardians) provided voluntary written informed consent.

Exclusion Criteria:

* Known allergy to local anesthetic agents.
* Presence of infection or skin disease at the planned puncture site.
* Severe coagulation disorders or current use of anticoagulant medications that cannot be safely discontinued for the procedure.
* Presence of severe cardiopulmonary or neurological disease.
* Inability to cooperate with regional or general anesthesia.
* Pregnancy or lactation.
* Presence of severe psychiatric illness or cognitive impairment that would hinder participation.
* Long-term use of analgesic medications.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale(NRS) | At baseline (before therapy),At 2hours post-surgery, At 6hours post-surgery、At 12hours post-surgery、At 24hours post-surgery.
  The NRS, Numerical Rating Scale, is a rating system from 0 to 10, where 0 represents "no pain" and 10 represents the worst possible pain.

SECONDARY OUTCOMES:
Total Postoperative Analgesic Consumption | At 24 hours post-surgery.
  The total amount of analgesic medication (including opioids and non-opioids, converted to morphine equivalents if necessary) used by patients from the end of surgery up to 24 hours post-surgery.
Postoperative Nausea and Vomiting (PONV) | At 24 hours after surgery
  The incidence and severity of nausea and vomiting experienced by patients after surgery.
Patient Satisfaction Score | At 24 hours after surgery
  Patient satisfaction with postoperative analgesia was assessed using a structured satisfaction survey. This survey employed a 10-point numerical rating scale, where 0 indicated complete dissatisfaction and 10 represented the highest level of satisfaction. The survey instrument encompassed evaluations of several key dimensions, including pain control, comfort, and the level of trust in the medical team.
Postoperative Recovery Status | From the end of anesthesia up to 24 hours post-surgery.
  Assessment of patient recovery status, including consciousness level, respiratory status, circulatory status, and overall well-being after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyu Wang, MM, Principal Investigator — Inner Mongolia Baogang Hospital
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2026-January 2031
Access Criteria: A proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed.